CLINICAL TRIAL: NCT04352660
Title: Subconjunctival Versus Direct Scleral Application of Mitomycin-C in Trabeculectomy
Brief Title: Subconjunctival Versus Direct Mitomycin C in Trabeculectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jiun Do, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 151621
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Open Angle Glaucoma
Keywords: trabeculectomy, mitomycin-C, glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Mitomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injection group (Active Comparator): MMC delivered by preoperative subconjunctival injection
  Interventions: Drug: Mitomycin-C injection
- Sponge group (Active Comparator): MMC delivered by intraoperative direct scleral application with impregnated cellulose sponges
  Interventions: Drug: Mitomycin-C sponge

INTERVENTIONS:
Drug: Mitomycin-C injection — MMC delivered by preoperative subconjunctival injection
  Arms: Injection group
Drug: Mitomycin-C sponge — MMC delivered by intraoperative direct scleral application with impregnated cellulose sponges
  Arms: Sponge group

SUMMARY:
Trabeculectomy is routinely used as a surgical treatment for open angle glaucoma. Success of trabeculectomy is greatly augmented by the use of antimetabolites to inhibit wound healing, specifically Mitomycin C (MMC). MMC can be applied to the eye at various sites, concentrations and times. This study aims to compare the two application routes that are commonly employed: subconjunctival pre-operative injection and intraoperative direct scleral application in terms of IOP lowering effect, bleb appearance and complications.

DETAILED DESCRIPTION:
Trabeculectomy is widely used as a surgical treatment of uncontrolled open glaucoma. Success of trabeculectomy at halting or slowing glaucoma progression primarily relies on the extent of conjunctival and sclera wound healing. The success rates of trabeculectomy increased dramatically with the introduction of anti-metabolites. For more than two decades mitomycin-c (MMC), a chemotherapeutic agent capable of decreasing fibroblast activity and modulating wound healing at the bleb, has been used with trabeculectomy. The complications of MMC are well known and several studies have described various methods of application based on exposure time, dose and surface area. Numerous retrospective and prospective studies have compared the efficacy of MMC applied beneath the conjunctival flap with soaked sponges versus intrascleral application. In 2008, Lee et al. first described an alternative route of application: subconjunctival injection of MMC directly into the intra-Tenon area. Seventy-six eyes with primary and secondary open angle glaucoma underwent trabeculectomy with this approach and were followed for one year post-operatively. Eighty-six percent of eyes achieved an IOP <21 mm Hg and 57% an IOP<14 mm Hg at one year without adjunctive drops. Transient complications included hyphema, bleb leak and choroidal detachment. The advantages of injected MMC are primarily in controlling the exact dosage and area of application and reduced surgical time. Lim et al. retrospectively reviewed the outcomes of trabeculectomy in 57 eyes using sponge application directly to the sclera versus intra-tenon injection. IOP was significantly lower in the injection group at 1 month, 1, 2, and 3 years. Trabeculectomy success (IOP<21mm Hg or IOP >20% below baseline without medications or additional surgery) was greater in the injection group at 3 years. The sponge group experienced more encapsulated blebs but complication rates were similar in both groups. To date, there have been no prospective studies comparing the IOP-lowering efficacy and safety of intra-tenon injection versus direct scleral application of MMC.

ELIGIBILITY:
Inclusion Criteria:

* medically uncontrolled glaucoma
* healthy and freely mobile conjunctiva in superior bulbar region

Exclusion Criteria:

* previous incisional glaucoma surgery
* no light perception vision
* pregnant or nursing women
* iris neovascularization or proliferative retinopathy
* iridocorneal endothelial syndrome
* chronic or recurrent uveitis
* steroid-induced glaucoma
* pathologic myopia or refractive error less than -6.00 diopters
* unwillingness or inability to give consent
* inability to return for scheduled protocol visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiun L Do, MD, PhD, Principal Investigator — UCSD; Robert N Weinreb, MD, Principal Investigator — UCSD; Benjamin Xu, MD, PhD, Principal Investigator — UCSD

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Injection Group | Sponge Group
Started | 50 | 50
Completed | 36 | 40
Not Completed | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Injection Group | Sponge Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (13.4) | 74.2 (9.5) | 72.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 24 | 26 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 28 | 55
  Asian | 9 | 7 | 16
  Hispanic | 9 | 5 | 14
  Black | 2 | 3 | 5
  Other | 3 | 7 | 10
Diagnosis [Count of Participants; unit: Participants]
  Primary open angle glaucoma | 45 | 43 | 88
  Pseudoexfoliation glaucoma | 2 | 3 | 5
  Pigmentary glaucoma | 0 | 1 | 1
  Chronic angle closure glaucoma | 1 | 0 | 1
  Other | 2 | 3 | 5
Visual Acuity [Mean (Standard Deviation); unit: logMAR] | 0.31 (0.34) | 0.36 (0.52) | 0.335 (0.44)
Preoperative Visual Field Mean Deviation [Mean (Standard Deviation); unit: decibels] — Visual field mean deviation is measured in decibels (dB) and is the amount of visual field loss compared to age matched controls (people with no eye diseases or visual field loss). The brightness of flashes of light is measured in decibels and used to test the peripheral visual field. Subjects able to see dimmer lights than age matched controls will have positive values. Subjects who require brighter stimuli than age matched controls will have negative values.
  decibels | -17.19 (7.90) | -15.87 (8.09) | -16.53 (8.00)
Preoperative Pattern Standard Deviation [Mean (Standard Deviation); unit: decibels] — Visual field pattern standard deviation is measured in decibels (dB) and is the amount of irregular visual field loss compared to age matched controls (people with no eye diseases or visual field loss). The absolute values of the difference between visual field threshold value and the average visual field sensitivity are summed. Subjects with focal visual field defects will have a large pattern standard deviation. Subjects with normal or diffuse visual field defects will have a small pattern standard deviation.
  decibels | 9.4 (3.6) | 8.9 (3.2) | 9.15 (3.40)
Preoperative Intraocular Pressure [Mean (Standard Deviation); unit: mm Hg] — Intraocular pressure is measured in millimeters of mercury . The intraocular pressure is measured in subjects using Goldmann applanation tonometry.
  mm Hg | 21.1 (7.2) | 21.8 (9.3) | 21.45 (8.3)
IOP Goal [Mean (Standard Deviation); unit: mm Hg] | 11.8 (0.9) | 12.7 (2.2) | 12.2 (1.7)
Number of Medications [Count of Participants; unit: Participants]
  None | 0 | 4 | 4
  1 | 4 | 6 | 10
  2 | 6 | 12 | 18
  3 | 21 | 21 | 42
  4 | 17 | 7 | 24
  5 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Intraocular Pressure Reduction Thresholds
Description: Percentage of patients achieving at least a 30% mean intraocular pressure reductions from baseline and with an intraocular pressure <21 mm Hg. Subjects that met this criteria without the use of intraocular pressure lowering medications were classified as "Complete Success." Subjects that met this criteria but required the use of intraocular pressure lowering medications were classified as "Qualified Success." Subjects that failed to meet this criteria were classified as "Failure." Subjects that failed to meet this criteria and required additional glaucoma surgery were classified as "Complete Failure."
Time Frame: 6 months
Population: 14 subjects in the Injection group were lost to follow up at the 6 month postoperative visit. 10 subjects from the Sponge group were lost to follow up at the 6 month postoperative visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Injection Group | Sponge Group
Number analyzed (Participants) | 36 | 40
Participants
  Complete Success | 21 | 21
  Qualified Success | 1 | 3
  Failure | 6 | 9
  Complete Failure | 8 | 7

2. Secondary Outcome: Bleb Morphology
Description: Bleb morphology at 6 months was graded using Indiana Bleb Appearance Grading Scale. Bleb height was graded on a scale of 0 to 3 (0: flat bleb without visible elevation, 1: low bleb elevation, 2: moderate bleb elevation, 3: high bleb elevation). Bleb extent was graded on a scale of 0 to 3 (0: no visible bleb extent to less than 1 clock hour, 1: extent equal to or greater than 1 clock hour but less than 2 clock hours, 2: extent equal to or greater than 2 clock hours but less than 4 clock hours, 3: extent equal to or greater than 4 clock hours). Bleb vascularity was graded on a scale of 0 to 4 (0: avascular/white, 1: avascular/cystic, 2: mild vascularity, 3: moderate vascularity, 4: extensive vascularity). Scales are descriptive and do not necessarily represent better or worse outcomes.
Time Frame: 6 months
Population: In the injection group, 14 subjects were lost to follow up and 17 subjects did not undergo bleb assessments at 6 months.In the sponge group, 10 subjects were lost to follow up and 20 subjects did not undergo bleb assessments at 6 months.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Injection Group | Sponge Group
Number analyzed (Participants) | 19 | 20
scores on a scale
  Height | 1.6 [1.3 to 1.9] | 1.7 [1.4 to 1.9]
  Extent | 2.2 [1.9 to 2.5] | 2.0 [1.7 to 2.3]
  Vascularity | 1.5 [1.2 to 1.9] | 1.5 [1.2 to 1.8]

3. Secondary Outcome: Medications
Description: Number of intraocular pressure lowering medications used by the patient at follow up visit.
Time Frame: 6 months
Population: In the injection group, 14 subjects were lost to follow up and 1 subject did not have medications documented at 6 months. In the sponge group, 10 subjects were lost to follow up and 2 subjects did not have medications documented at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Injection Group | Sponge Group
Number analyzed (Participants) | 35 | 38
Participants
  0 | 30 | 32
  1 | 3 | 4
  2 | 1 | 1
  3 | 1 | 1

4. Secondary Outcome: Visual Acuity
Description: Change in visual acuity from baseline
Time Frame: 6 months
Population: In the injection group, 14 subjects were lost to follow up at 6 months. In the sponge group, 10 subjects were lost to follow up at 6 months.
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Injection Group | Sponge Group
Number analyzed (Participants) | 36 | 40
logMAR | 0.11 [0 to 0.22] | 0.03 [-0.09 to 0.14]

5. Secondary Outcome: Number of Participants With Surgical Complications
Description: Number of eyes that experienced surgical complications following surgery
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Injection Group | Sponge Group
Number analyzed (Participants) | 50 | 50
participants
  Hypotony Maculopathy | 3 | 1
  Choroidal Effusions | 2 | 5

6. Secondary Outcome: Number of Participants Requiring Additional Surgery
Description: Number of eyes requiring additional surgery from each group
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Injection Group | Sponge Group
Number analyzed (Participants) | 50 | 50
participants
  Trab Revision | 8 | 5
  GDD | 2 | 1
  Xen | 0 | 1
  Trabectome | 0 | 1
  Any Surgery | 8 | 7
  CEIOL | 8 | 5
  YAG | 0 | 1

7. Secondary Outcome: Postoperative Interventions
Description: Mean number of postoperative interventions (needling, antifibrotic injections) performed in each group
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: number of procedures
Arm/Group | Injection Group | Sponge Group
Number analyzed (Participants) | 50 | 50
number of procedures
  5FU Injection | 3.3 [2.6 to 4.0] | 3.2 [2.2 to 4.3]
  Laser suture lysis | 2.0 [1.5 to 2.5] | 1.6 [1.1 to 2.1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Injection Group | Sponge Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 5/50 | 6/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Injection Group (N=50) | Sponge Group (N=50)
Hypotony maculopathy (Eye disorders) | 3 | 1
Choroidal effusions (Eye disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT04352660/Prot_SAP_000.pdf